CLINICAL TRIAL: NCT04223947
Title: Endoscopic Characterization of Colorectal Neoplasia With the Different Published Classifications: a Prospective Comparative Study Involving Gastroenterologists From Trainees to Experts
Brief Title: Endoscopic Characterization of Colorectal Neoplasia With the Different Published Classifications: a Prospective Comparative Study
Status: Completed | Type: Observational
Sponsor: Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Jean Christophe Saurin, Professor, Hôpital Edouard Herriot
Other Study IDs: SFED2
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: ENDOSCOPIC CHARACTERIZATION
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: DIGESTIVE ENDOSCOPY — DIGESTIVE ENDOSCOPY

SUMMARY:
Endoscopic characterization of colorectal lesions has become essential to predict histology and choose the best therapeutic strategy. We have created the CONECCT classification grouping all the endoscopic criteria already published in a single table. To validate this classification, we carried out this comparative study evaluating the endoscopic characterization performance of all recognized classifications and CONECCT in terms of inter-observer agreement and histological prediction.

ELIGIBILITY:
Inclusion Criteria:

* none

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal lesions
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of inter observer agreement in the use of current endoscopic classifications | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- hôpital Edouard Herriot, Lyon, Auvergne-Rhône-Alpes, France